CLINICAL TRIAL: NCT05974241
Title: Irritability in Children With ADHD and Emotion Dysregulation: Clinical Profiles, Neuropsychological Characteristics , and Pharmacological Treatment: A Cross-over Study
Brief Title: Irritability in Children With ADHD and Emotion Dysregulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chin-Bin Yeh, MD, PhD, Attending Physician, Tri-Service General Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSGH-C106-103
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Irritable Mood; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Aripiprazole

STUDY DESIGN:
Intervention Model Description: A three-step, open-label, 10 week pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacological treatment (Experimental): During the first step, the subjects received pharmacological treatment of methylphenidate with flexible dosage for 4 weeks. Those subjects who had suboptimal response to methylphenidate entered the second step with aripiprazole. After 4 weeks of treatment, those had suboptimal response to aripiprazole entered the third step and received the treatment of combination of methylphenidate and aripiprazole for two weeks (3rd step).
  Interventions: Drug: Methylphenidate, aripiprazole, and combination

INTERVENTIONS:
Drug: Methylphenidate, aripiprazole, and combination — Methylphenidate (4 weeks), aripiprazole (4 weeks), and the combination (2weeks). The primary outcome was improvement of irritability as measured by Aberrant Behavior Checklist-irritability subscale (ABC-I). During the first step, the subjects received pharmacological treatment of methylphenidate with flexible dosage for 4 weeks. Those subjects who had suboptimal response to methylphenidate (reduction of ABC-I score < 25%) entered the second step and the medication was switched to aripiprazole. After 4 weeks of treatment, those whose ABC-I scores reduced < 25% entered the third step and received the treatment of combination of methylphenidate and aripiprazole for two weeks (3rd step).
  Other Names: Ritalin/Concerta, Abilify, and combination

SUMMARY:
Objective:

Emotion dysregulation is common among children with ADHD and associated with a broad range of adult psychopathology, which is similar to the longitudinal outcomes of childhood irritability. However, the profiles of irritability in children with ADHD and emotion dysregulation has been understudied. This study aimed to investigate the efficacy of methylphenidate and aripiprazole in the treatment of irritability in children with ADHD and emotion dysregulation. In addition, the clinical profiles and neuropsychological characteristics of irritability in children with ADHD were explored.

DETAILED DESCRIPTION:
Methods:

A three-step, open-label, 10 week pilot study was conducted. Methylphenidate (4 weeks), aripiprazole (4 weeks), and the combination (2weeks) were examined in sequence as the treatment for irritability in children with ADHD and emotion dysregulation, defined by the CBCL-Dysregulation Profile. The primary outcome was improvement of irritability as measured by Aberrant Behavior Checklist-irritability subscale (ABC-I). During the first step, the subjects received pharmacological treatment of methylphenidate with flexible dosage for 4 weeks. Those subjects who had suboptimal response to methylphenidate (reduction of ABC-I score < 25%) entered the second step and the medication was switched to aripiprazole. After 4 weeks of treatment, those whose ABC-I scores reduced < 25% entered the third step and received the treatment of combination of methylphenidate and aripiprazole for two weeks (3rd step).

Clinical profiles of irritability were evaluated with the Affective Reactivity Index (ARI), the Strengths and Difficulties Questionnaire, the Social Adjustment Inventory for Children and Adolescents, and the Autism Behavior Checklist-Taiwan Version. The neurophysiological characteristics of the subjects were assessed by three Cantab subtests: Emotion Recognition Task, One Touch Stockings of Cambridge, and Spatial Working Memory. The aforementioned measurements were administered at baseline and at the end of each step.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 to 18 who have ADHD and emotion dysregulation, defined by the CBCL-Dysregulation Profile.

Exclusion Criteria:

* Patients who are not willing to participate in the study after detailed explanation.
* Patients who have intellectual disability or could not follow the investigator's instructions.
* Patients who have severe neurological or mental illness like epileptic disorder, schizophrenia, bipolar disorder, or uncontrolled suicide risk.
* Patients who have severe medical illness or surgical conditions like uncontrolled abnormal thyroid function, or severe congenital heart disease.
* Patients who are allergic to methylphenidate or aripiprazole.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-irritability subscale (ABC-I) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  The ABC is an instrument developed to assess emotional and behavioral difficulties in individuals with developmental disabilities. However, its irritability subscale (ABC-I) is a proven well-validated and widely used rating inventory for measuring irritability in neurotypical children. This subscale consists of 15 items about irritability, aggression, tantrums, agitation, and unstable mood.

SECONDARY OUTCOMES:
Affective Reactivity Index (ARI) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  The ARI was created as a dimensional measurement of irritability with both parent-report and self-report form. This questionnaire, assessing for symptoms of irritability in the previous 6 months, is composed of 6 items, and the 7th item on functional impairment is rated on a three-point scale (ranging from 0 for "not true" to 2 for "certainly true"). The reliability and validity of the ARI in typically developed children has been previously reported. The sum of scores of the first six items was used in this present study.
Social Adjustment Inventory for Children and Adolescents (SAICA) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  The SAICA was designed for children and adolescents aged 6-18 years, and provided a systematic evaluation of children's and adolescents' adaptive functioning. It assessed social adjustment in four major role areas: school, spare-time activities, peer relations, and home life. The scoring of each item ranges from 1 for positive/not a problem, to 4 for negative/severe problem. The children or adolescents with higher scores had either poorer functioning or more severe problems in the assessed domain.
The Strengths and Difficulties Questionnaire (SDQ) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  The SDQ is a questionnaire for assessing the psychological problems and strengths in children, consisting of 25 items categorized as 5 subscales based on factor analyses: emotional symptoms, conduct problems, hyperactivity, peer problems, and prosocial behavior. An impact supplement added to the SDQ provides additional information on the target child's possible difficulties and the burden for others. Previous studies report that the Chinese version of the SDQ is a reliable and valid instrument for clinical studies in Taiwan.
Cantab subtest-- Emotion Recognition Task (ERT) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  The outcome measures for ERT cover percentage and number correct or incorrect and overall response latencies, which can be looked at either across individual emotions or across all emotions at once.
Cantab subtest-- One Touch Stockings of Cambridge (OTS) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  Outcome measures include the number of problems solved on first choice, mean choices to correct, mean latency (speed of response) to first choice and mean latency to correct. Each of these measures may be calculated for all problems, or for problems with a specified number of moves (one-move to five or six moves).
Cantab subtest-- Spatial Working Memory (SWM) | 4 weeks for the 1st step, 4 weeks for the 2nd step, and 2 weeks for the 3rd step
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token) and strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Bin Yeh, MD., PhD., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

REFERENCES:
- [Derived] Pan PY, Yeh CB. The Role of Methylphenidate and Aripiprazole in the Treatment of Emotion Dysregulation in Children With ADHD. J Clin Psychopharmacol. 2025 Jul-Aug 01;45(4):356-363. doi: 10.1097/JCP.0000000000002002. Epub 2025 Apr 16. PMID 40238929